CLINICAL TRIAL: NCT04754243
Title: A Higher Ovulation and Pregnancy Rates in Patients With Unexplained Infertility After Application of ANTIUI Protocol: A Randomized Multicenter Controlled Study
Brief Title: New Protocol in Unexplained Infertility
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Assistant professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANTIUI
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Unexplained Infertility
MeSH Terms: interventions — Gonadotropins

STUDY DESIGN:
Intervention Model Description: 2 parallel groups each is receiving different intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Will receive ANTIUI protocol
  Interventions: Drug: Gonadotropin
- Control group (Active Comparator): Will receive standard protocol in IUI and unexplained infertility
  Interventions: Drug: Standard protocol in IUI

INTERVENTIONS:
Drug: Gonadotropin — Giving patients gonadotropins and antagonist cetrotide
  Arms: Study group
Drug: Standard protocol in IUI — Giving patients gonadotropins without antagonist cetrotide
  Arms: Control group

SUMMARY:
The new protocol ANTIUI provides good results regarding ovulation and pregnancy rates in patients with unexplained infertility

DETAILED DESCRIPTION:
Patients with unexplained infertility has normal investigations regarding hormonal, structural data. Semen is normal but no pregnancy occurs.

Before trying ICSI, we could help these patients with ANTIUI

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertility
* Duration less than 5 years
* Good ovarian reserve AMH> 1.1
* Normal patent tubes
* No previous trials of IUI with the same protocol

Exclusion Criteria:

* Age > 35 years
* Duration of infertility> 5 years
* Abnormal semen
* Hypoplastic tubes
* prior failed ICSI

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ovulation | 6 months
  Disappearance of mature follicle
Pregnancy | 6 months
  Number of pregnant cases

CONTACTS AND LOCATIONS:
Locations (1):
- Ayman Shehata Dawood, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Within 6 MONTHS
Supporting Information: Study Protocol
Time Frame: 6 months